CLINICAL TRIAL: NCT06181344
Title: Implementation and Evaluation of a Fear of Cancer Recurrence Screening, Referral and Management Program for Chinese Cancer Survivors: a Stepped Wedge and Cluster Randomized Trial
Brief Title: Implementation and Evaluation of a Fear of Cancer Recurrence Screening, Referral and Management Program
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Health and Medical Research Fund (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: UW23-458
Record Dates: First submitted 2023-12-12; First posted 2023-12-26 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Fear of Cancer Recurrence; Cancer
Keywords: implementation study; Screening and referral program
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: This study will use a stepped wedge cluster randomized controlled trial design in which the intervention is introduced stepwise across study units. After obtaining the consent form from the five clinical care units, they will be randomized to one of the two roll-out schedules with a 4-month duration each. All the study units will start the trial in a control condition (i.e., no implementation strategies used), then sequentially cross over from the control condition to the intervention condition, until all sites are receiving the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- implementation condition (Experimental): Under implementation condition, a fear of cancer recurrence screening program will be implemented in routine oncological clinics using 5 implementation strategies including training, audit and feedback, facilitation and adaptable workflow.
  Interventions: Behavioral: FCR screening and referral program
- Control condition (No Intervention): In the control condition, the clinical outpatient operation is performed as usual. The FCR screening tool and referral forms will be provided to the study sites and nursing staff are encouraged to adopt fear of cancer recurrence screening. Patients referred to JCICC will be managed following the predefined clinical pathway triage system. A briefing session about the purpose of the implementation program and the introduction of the FCR screening tool will be given to the staff at each study unit before the start of the first 4-months control condition. The briefing session will be recorded for the purpose of fidelity assessment.

INTERVENTIONS:
Behavioral: FCR screening and referral program — Five implementation strategies will be conducted individually for each of the study unit at the timepoint when the study unit is being randomly allocated to the implementation condition. For each study unit, all nurses will first receive a half-day training. Each study unit under the implementation condition will receive weekly audit and feedback reports to summarize the proportion of eligible patients, proportion of eligible patients being screened, proportion of patients appropriately referred to JCICC. The senior research assistant with a nursing background will receive training and mentoring from the PI and will be the guided facilitator. The guided facilitator will conduct weekly site visits to address operational issues arise during the implementation. Lastly, while the choice of symptom assessment tool and referral criteria are standardized and cannot be modified, the routine workflow for each study unit can be adjusted according to its context and resources.
  Arms: implementation condition

SUMMARY:
The purpose of this study is to evaluate the process and outcomes of an implementation program designed to implement fear of cancer screening, referral and management into routine cancer care clinics, using a stepped-wedge cluster randomized controlled trial.

DETAILED DESCRIPTION:
This study aims to test if a systematic fear of cancer screening program that employs implementation strategies including training, reflecting, evaluating, facilitating and adapting, increases the proportion of eligible patients screened and referred compared to usual control with no implantation strategies used. This study hypothesize that the implementation program will increase (i) the proportion of eligible patients screened and (ii) the proportion of patients with high fear of cancer referred for psychosocial support. For process evaluation, this study aims to use qualitative methods to assess the patients' and service providers' experience of the implementation program, and identify contextual factors (e.g., potential barriers and facilitators) likely to influence its adoption, implementation, and sustainability.

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed with non-metastatic breast, gynecological, or colorectal cancer, and who have completed primary and adjuvant treatment within the past two years will be eligible for the proposed screening program.

Exclusion Criteria:

* All cancer patients beyond two years post-treatment; and diagnosed with metastatic cancer or non-breast, non-gynecological, and non-colorectal cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1980 (Estimated)
Dates: Start 2024-07-26 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in the number of eligible patient screened | Pre- and post-implementation phase, up to 24 months
  The primary outcome (the measurement of the reach) is the changes in the number of eligible patients screened. Using a standardized reporting form, each study site will be asked to submit a weekly record of a total number of eligible patients per clinic and the number of patients screened.
Change in the number of eligible patient referred | Pre- and post-implementation phase, up to 24 months
  The primary outcome (the measurement of the reach) is the changes in the number of eligible patients referred based on the predefined scores. Using a standardized reporting form, each study site will be asked to submit a weekly record of a total number of eligible patients per clinic and the number of patients referred.

SECONDARY OUTCOMES:
Change in referral uptake | Pre- and post-implementation phase, up to 24 months
  The secondary outcome is the change in uptake of the referral, i.e. the proportion of referred patients accepting services.
Process evaluation in providers by conducting qualitative interviews | Pre- and post-implementation phase, up to 24 months
  Using qualitative approach with service providers (i.e. the nurses) to identify facilitators and barriers for the implementation of the symptom distress screening program, as well as their overall experience. All nursing staff from the study units involved in the symptom distress screening will be invited to join the qualitative study at the post-implementation phase.
Process evaluation in patients by conducting qualitative interviews | Pre- and post-implementation phase, up to 24 months
  The investigators will also conduct qualitative interviews to explore patients' experiences with symptom distress screening and referral if appropriate. Patients who are referred for support services will be approached by the research assistant who will explain the purpose of the study and nature of participation, with an emphasis on confidentiality and anonymity. If agreeing to participate, the RA will obtain a written consent and each subject will subsequently participate in in-depth interview by a trained interviewer. For patients who decline to be referred for support services, the investigators will ask the nursing staff to invite the patients to join the qualitative study. The investigators will recruit patients from both implementation and control conditions as it will enable us to compare patients' experience.
Number of staff receiving training | Pre- and post-implementation phase, up to 24 months
  All nurses will first receive a half-day training on how to administer the symptom distress screening tool, evaluate patients' reported symptom distress, refer patients to and follow-up for referred patients. The investigators will record the number of invited staff attending the half-day training workshop.
Change in staff knowledge about the implementation of the screening programme assessed using categorical Likert scales | Pre- and post-implementation phase, up to 24 months
  The investigators will assess the staff knowledge at pre- and post-training workshop and again at the end of the implementation study using a 6 points-categorical Likert scale (0-5) for participants' knowledge about the implementation of the screening program. Such information will be served as implementation indicators to facilitate the interpretation of the study findings.
Change in staff's belief in the symptom distress screening programme assessed using categorical Likert scales | Pre- and post-implementation phase, up to 24 months
  The investigators will assess the staff's belief at pre- and post-training workshop and again at the end of the implementation study using a 6 points-categorical Likert scale (0-5) for participants' beliefs towards the symptom distress screening programme. Such information will be served as implementation indicators to facilitate the interpretation of the study findings.
Change in staff self-efficacy in administrating the symptom distress screening programme assessed using categorical Likert scales | Pre- and post-implementation phase, up to 24 months
  The investigators will assess the staff's self-efficacy at pre- and post-training workshop and again at the end of the implementation study using a 6 points-categorical Likert scale (0-5). Such information will be served as implementation indicators to facilitate the interpretation of the study findings.

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Ng, PhD, Principal Investigator — The University of Hong Kong
Locations (2):
- Hong Kong (2):
  - KWH Breast clinic, Hong Kong
  - QMH department of Surgery, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be available from the PI upon reasonable reques
Supporting Information: Study Protocol
Time Frame: Starting 6 months after publication
Access Criteria: Information will be available from the PI upon reasonable request. The author to review requests is the PI.